CLINICAL TRIAL: NCT00887081
Title: Phase IV Study of Effectiveness of Interferon and Ribavirin Treatment in Thalassemia Major Patients With Chronic Viral Hepatitis C
Brief Title: Interferon and Ribavirin Treatment in Patients With Hemoglobinopathies
Acronym: IFNRIBAHE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera V. Cervello (Other)
Responsible Party: Aurelio Maggio, M.D., Azienda Ospedaliera V. Cervello
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AOVCervello1
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Hemoglobinopathies
Keywords: antiviral treatment in hemoglobinopathies; management of chronic viral hepatitis C infection; antiviral treatment
MeSH Terms: conditions — Hemoglobinopathies | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interferon and Ribavirin (Experimental): Patients with hemoglobinopathy will receive Interferon and Ribavirin
  Interventions: Drug: PEG-IFN alpha2a or PEG-IFN alpha2b and Ribavirin

INTERVENTIONS:
Drug: PEG-IFN alpha2a or PEG-IFN alpha2b and Ribavirin — PEG-IFN alpha2a 180 mcg weekly or PEG-IFN alpha2b 1.5 mcg/kg of body weight weekly plus ribavirin 800-1200 mg daily according to body weight.
  Other Names: Pegasis; Rebetol

SUMMARY:
Worldwide, several studies report that 4.4% to 85.4% of thalassemia patients were positive for anti hepatitis C antibodies. Recently, three different studies reported the efficacy and the safety of combination therapy with pegylated interferon and ribavirin in thalassemic patients. This study is carried ahead to assess the impact of combination therapy with pegylated-interferon and ribavirin in a large cohort of italian patients with beta thalassemia major - transfused and not transfused, sickle cell disease and sickle/beta-thalassemia.

DETAILED DESCRIPTION:
Infection is more common in patients who received a high number of blood transfusions before 1990. The prevalence of HCV infection is higher in Italy, where more than 70% of thalassemia major patients are HCV-RNA positive. In Italy and worldwide, genotype 1 is the most frequent. Regarding the prevalence of cirrhosis, the clinical data of different cohorts of thalassemia patients showed a rate of cirrhosis ranging from 10% to 20%. Male sex, high serum ALT values, and a positive serum test for qualitative HCV-RNA are significantly associated with severe fibrosis or cirrhosis. Cirrhosis related to hepatitis C virus infection is the major risk factor for development of hepatocellular carcinoma and is a major cause of liver failure. An Italian study that reported clinical data of 22 thalassemia patients with hepatocellular carcinoma concluded that the development of hepatocellular carcinoma is associated with the presence of cirrhosis, male gender, age over 35 years, and active HCV infection. Another prospective study reported a 2% incidence of new HCC during the follow-up of 105 adult thalassemia patients cohort. Yet before 2000, several controlled trials reported that combination therapy with alpha-interferon, given three times a week, and ribavirin, given every day, was more effective than interferon alone.Recently, three different studies reported the efficacy and the safety of combination therapy with pegylated interferon and ribavirin in thalassemic patients. Less extensive data are present actually in literature about efficacy of combination therapy with pegylated interferon and ribavirin in HCV infected patients with sickle cell disease or sickle/beta-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia Major or Sickle Cell Disease or Sickle/Beta Thalassemia patients
* Regularly transfused (hemoglobin ≥ 9.5 gr/dl) or not transfused, under or not iron chelation regimen
* With positivity to HCV-RNA and chronic liver disease with or without cirrhosis, naïve or non-responder or relapser after interferon mono-therapy

Exclusion Criteria:

* Thalassemia Major or Sickle Cell Disease or Sickle/Beta Thalassemia patients with not compensated liver failure or heart failure
* Low white blood cells (neutrophils < 1.500/mmc and/or white blood cells < 3.000/mmc)
* Low platelets count (< 100.000/mmc)
* Significant positivity to Coombs test with clinical and serologic evidence of immune hemolytic anemia, severe endocrinopathy, detection of high titre autoantibodies, co-infection with HBV (HbsAg positive)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
A sustained virological response (SVR), defined as absence of HCV RNA in serum by a highly sensitive test at the end of treatment and 6 months late. | from 6 to 12 months

SECONDARY OUTCOMES:
Early virological response (EVR) , defined as the loss of HCV RNA during the first 12 weeks of therapy; main side effects enclosing changes in blood transfusion requirement; increase in ferritin levels and variations in chelation treatment | from 6 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Maggio, M.D., Study Chair — Azienda Ospedaliera V. Cervello; Gaetano Restivo, M.D., Principal Investigator — Azienda Ospedaliera V. Cervello; Disma Renda, M.D., Study Director — Azienda Ospedaliera V. Cervello
Locations (1):
- AOVCervello, Palermo, Italy